CLINICAL TRIAL: NCT05090176
Title: Title: Povidone-soaked Sutures Versus Ordinary Sutures for Reducing Surgical Site Infection: Randomize Control Trial Study in General Surgery Cases of Hospital Universiti Sains Malaysia
Brief Title: Title: Povidone-soaked Sutures Versus Ordinary Sutures for Reducing Surgical Site Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, SITI HAFZAN, Principle investigator, Universiti Sains Malaysia
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: fz03
Record Dates: First submitted 2021-09-14; First posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Efficacy Povidone Soaked Suture in Reducing Surgical Site Infection
Keywords: suture; povidone; surgical site infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: randomized control trial, double blind
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- povidone-soaked suture (Experimental): The patient is randomized, those with povidone-soaked suture group will be prepared for povidone-soaked suture during wound closure.
  The absorbable suture will be soaked into povidone for 3 mins before the wound closure.
  Interventions: Other: povidone-soaked suture
- ordinary suture (Active Comparator): the patient is randomized, those with ordinary suture group will proceed with wound closure as usual manner following the standard practice.
  Interventions: Other: ordinary suture

INTERVENTIONS:
Other: povidone-soaked suture — suture soak with povidone solution for 3 mins
  Arms: povidone-soaked suture
Other: ordinary suture — suture no need to soak with povidone solution
  Arms: ordinary suture

SUMMARY:
To determine efficacy of using 3 minutes povidone-soaked suture in reducing surgical site infection during wound closure in elective surgery.

DETAILED DESCRIPTION:
Participant recruitment and randomisation based on eligibility based on CONSORT.

Patient will get either package A or B which determine whether they are getting povidone-soaked suture or ordinary suture during wound closure.

Postoperative, follow up on D10 and D30 of patient well being and signs and symptoms of surgical site infection

ELIGIBILITY:
Inclusion Criteria:

* Age more than 12 years old
* Clean surgery or Clean- contaminated surgery
* Elective surgery

Exclusion Criteria:

* Age less than 12 years old
* Contaminated wound
* Dirty wound
* Allergy to povidone-iodine
* Pregnant
* Laparoscopic
* Emergency surgery

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-11-02 (Estimated)

PRIMARY OUTCOMES:
Povidone-soaked Sutures versus Ordinary Sutures for Reducing Surgical Site Infection: Randomize Control Trial Study in General Surgery Cases of Hospital Universiti Sains Malaysia | 6 months
  There is difference of outcome using povidone-soaked suture and ordinary suture. In this study, our hypothesis the suture with povidone-soaked will reduce the SSIs rate during closure and it will be assessed on day 10 and day 30 post-operative.
  Few measurement are used in detection of SSI based on clinical and biochemical measurement such as signs of inflammation and total white cell count.

SECONDARY OUTCOMES:
Povidone-soaked Sutures versus Ordinary Sutures for Reducing Surgical Site Infection: Randomize Control Trial Study in General Surgery Cases of Hospital Universiti Sains Malaysia | 6 months
  There is association between povidone-soaked suture and ordinary suture in reducing surgical site infection. There is difference of outcome using povidone-soaked suture and ordinary suture. In this study, our hypothesis the suture with povidone-soaked will reduce the SSIs rate during closure and it will be assessed on day 10 and day 30 post-operative.
  Few measurement are used in detection of SSI based on clinical and biochemical measurement such as signs of inflammation and total white cell count.
Povidone-soaked Sutures versus Ordinary Sutures for Reducing Surgical Site Infection: Randomize Control Trial Study in General Surgery Cases of Hospital Universiti Sains Malaysia | 6 months
  There is difference in the extent of intervention needed to manage SSIs in wounds closed with povidone-soaked suture and ordinary suture.
  This hypothesis measure how far that the management of SSIs whether non-operative or operative treatment is needed.
  This is base on antibiotic use, dressing and surgical intervention such as debridement.

CONTACTS AND LOCATIONS:
Overall Officials: SITI HAFZAN ABD KARIM, MD, Principal Investigator — UNIVERSITI SAINS MALAYSIA- HEALTH CAMPUS
Locations (1):
- Universiti Sains Malaysia, Kubang Kerian, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: No